CLINICAL TRIAL: NCT02608515
Title: A Retrospective Chart Review Study of the Outcomes of Second Line Therapy With LEnalidomide/Dexamethasone in Greek Patients With Relapsed/Refractory Multiple MyEloma and the Treatment PatterNs Following Progressive Disease, "The LEGEND Study"
Brief Title: A Retrospective Chart Review Study of the Outcomes of 2nd Line Therapy With LEn/Dex in Greek Patients With R/R Multiple MyEloma and the Treatment PatterNs Following Progressive Disease
Acronym: LEGEND
Status: Completed | Type: Observational
Sponsor: Genesis Pharma S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: NIPMS-GENESIS-MM-GRC-002
Record Dates: First submitted 2015-11-17; First posted 2015-11-18 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
This non-interventional retrospective chart review study aims to evaluate the clinical outcomes of patients with RRMM receiving lenalidomide/dexamethasone (Len/Dex) treatment at 1st relapse and the treatment patterns following progressive disease as part of the routine clinical practice in Greece.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill ALL of the following criteria:

* Subjects of both genders, aged 18 years or older
* Subjects must have a relapsed or refractory MM diagnosis according to IMWG or EBMT criteria
* Subjects must have initiated second-line therapy with lenalidomide/dexamethasone according to the approved products' Summary of Product Characteristics (SmPC) between 01 January 2009 and 01 March 2014
* Subjects must have available medical files/records and detailed historical data on their disease course and clinical management
* Provision of signed ICF for collecting and analyzing medical data pertinent to the objectives of this study

Exclusion Criteria:

For the candidate subjects NONE of the following criteria should apply:

* Prior malignancy (within the 3 years preceding initial diagnosis of MM)
* Concurrent administration of anti-cancer regimens for malignancies other than MM between the time of initial MM diagnosis and time of second relapse
* Subject participation in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of approximately 220 patients with RRMM that started second-line treatment with lenalidomide/dexamethasone between 01 January 2009 to 01 March 2014 and who fulfill all study-specific eligibility criteria at the investigators' discretion will be included in this study
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the 12-month PFS rate in patients treated with Len/Dex at 1st relapse | 12 months
  PFS rate

CONTACTS AND LOCATIONS:
Overall Officials: Kiki Karvounis, Study Director — Medical Department of Genesis Pharma SA
Locations (1):
- Patra, Pátrai, Greece

REFERENCES:
- See also: Published Manuscript — https://link.springer.com/article/10.1007/s00277-018-3361-2